CLINICAL TRIAL: NCT00303147
Title: Cognitive and Health Benefits of Expressive Writing for Family Caregivers Under Stress
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Baycrest Centre for Geriatric Care (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11438
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2006-03-15 (Estimated); Status verified 2006-03

CONDITIONS: Stress, Psychological; Anxiety
Keywords: Expressive Writing; Written Emotional Expression; Caregiver Stress; Cognition
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Caregiver Burden

INTERVENTIONS:
Behavioral: Expressive Writing

SUMMARY:
The purpose of this study is to determine if expressive writing is an effective intervention for reducing stress, enhancing cognition, and improving quality of life for caregivers of older adults with dementia

DETAILED DESCRIPTION:
A significant and growing need exists to support caregivers of older adults with dementia, including methods of support that are easily implemented and targeted at caregivers who can not access multicomponent interventions. The current intervention examines the efficacy of one such approach: expressive writing (EW).

We are examining the efficacy of EW, in terms of its ability to reduce stress, enhance cognition, and improve well-being, by comparing it to two control conditions: objective writing about how caregivers spend their time (time management; TM) and objective writing about non-personal historical events (history writing; HW).

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver for an older adult with dementia
* Self-reported caregiver stress or burden
* Fluency in written/spoken English

Exclusion Criteria:

* non-family or non-primary caregiver
* existing use of expressive writing / diary

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-05; Study Completion 2005-07

PRIMARY OUTCOMES:
General Health Questionnaire
Impact of Events Scale
Zarit Burden Interview (short form)
California Verbal Learning Test
Ruff 2 & 7 Selective Attention Test
Wechsler Adult Intelligence Scale (WAIS)

CONTACTS AND LOCATIONS:
Overall Officials: Corey S Mackenzie, Ph.D., Principal Investigator — University of Toronto; Lynn Hasher, Ph.D., Principal Investigator — University of Toronto; David Goldstein, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada